CLINICAL TRIAL: NCT01824823
Title: A Randomized Placebo Controlled Phase II Trial of Afatinib (BIBW2992) as Adjuvant Therapy Following Chemoradiation in Patients With Head and Neck Squamous Cell Carcinoma at High Risk of Recurrence
Brief Title: Afatinib After Chemoradiation and Surgery in Treating Patients With Stage III-IV Squamous Cell Carcinoma of the Head and Neck at High-Risk of Recurrence
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E1311; NCI-2013-00357 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U10CA021115 (NIH)
Record Dates: First submitted 2013-04-02; First posted 2013-04-05 (Estimated); Results first posted 2016-04-04 (Estimated); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: afatinib; head and neck squamous cell carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Afatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (afatinib) (Experimental): Patients receive afatinib PO QD on days 1-28.
  Interventions: Drug: afatinib
- Arm B (placebo) (Placebo Comparator): Patients receive placebo PO QD on days 1-28.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: afatinib — Given PO
  Other Names: BIBW 2992
  Arms: Arm A (afatinib)
Other: placebo — Given PO
  Arms: Arm B (placebo)

SUMMARY:
This randomized phase II trial studies how well giving afatinib after chemoradiation and surgery works in treating patients with stage III-IV squamous cell carcinoma of the head and neck at high-risk of recurrence. Afatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Examine disease-free survival (DFS) given afatinib/placebo adjuvant therapy in patients with viable tumors in lymph nodes after neck dissection for suspected residual disease after concurrent chemoradiation.

SECONDARY OBJECTIVES:

I. Evaluate the recurrence rate, recurrence patterns, development of second primary malignancies, overall survival (OS) and toxicity of afatinib/placebo.

II. Evaluate on-target inhibition by afatinib, and determine circulating deoxyribonucleic acid (DNA) as a biomarker of afatinib resistance.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive afatinib orally (PO) once daily (QD) on days 1-28.

ARM B: Patients receive placebo PO QD on days 1-28.

In both Arms, treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 1 year and then every 12 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Patients must have pathological evidence of persistent primary and/or lymph node disease with viable tumor cells following primary concurrent chemoradiotherapy of locoregionally advanced (stage III/IV) HNSCC of the oral cavity, oropharynx, larynx, hypopharynx or p16-positive unknown primary of the head and neck region; persistent primary and/or lymph node disease with viable tumor cells will be determined by the histological determination of tumor viability defined as tumor cells with intact cellular compartments (i.e. cytoplasm and nucleus) that do not exhibit karyolysis, pyknosis, or karyorrhexis on haematoxylin and eosin (H&E) staining
* Patients must have undergone a neck dissection following completion of chemoradiotherapy and must have involved at the minimum a compartment dissection of nodal levels with residual abnormalities on post-treatment imaging studies and/or received a complete resection of the residual primary lesion with negative margins
* Patients must have achieved a complete response at the primary disease site after chemoradiotherapy or complete resection of the residual primary site disease with negative margins
* All persistent lymph node disease must have received at least 66 Gy of radiotherapy and must have been completely surgically resected prior to registration, and surgical incisions should be adequately healed
* Patients with extracapsular lymph node extension, perineural or lymphovascular invasion will be eligible
* Patients must be at least 6 weeks (42 days) and no more than 36 weeks (252 days) from completion of chemoradiation at the time of registration
* Patients will be eligible regardless of ability to swallow; patients with dysphagia may have afatinib/placebo administered via gastrostomy tube
* Absolute neutrophil count >= 1,000/mm^3
* Platelets >= 100,000/mm^3
* Total bilirubin =< 1.5 x the upper limit of normal (ULN)
* Aspartate amino transferase (AST) =< 3 x the ULN
* Alanine amino transferase (ALT) =< 3 x the ULN
* Calculated creatinine clearance must be >= 50 ml/min using the Cockcroft-Gault formula
* Prior cetuximab or any epidermal growth factor receptor (EGFR) inhibitors will not be permitted including cetuximab administered with a chemoradiotherapy or radiotherapy regimen
* As all patients in this study will have received prior full dose, curative-intent external-beam radiotherapy to the involved neck, no additional external-beam radiotherapy will be permitted prior to or during study participation
* Women of childbearing potential and sexually active males must be strongly advised to use an accepted and effective method of contraception
* Patients must have electrocardiogram (ECG) within 8 weeks prior to randomization to the study
* Patients must be assessed for cardiac function by echocardiogram (ECHO) or multi-gated acquisition scan (MUGA) within 8 weeks prior to randomization

Exclusion Criteria:

* Patients with known distant metastatic disease or with any gross residual disease following salvage primary tumor resection or neck dissection
* Known hypersensitivity to afatinib or any of the excipients of this product
* Prior adjuvant chemotherapy (aside from the initial induction chemotherapy followed by chemoradiotherapy or chemoradiotherapy regimen)
* History of acute myocardial infarction within 3 months prior to registration, and any history of uncontrolled angina, uncontrolled arrhythmia, or uncontrolled heart failure
* Pregnant or breast-feeding women
* Active infections, other cancers, or history of other cancers
* Participation in any other clinical trials or taking any other experimental medications
* Left ventricular dysfunction
* Evidence of interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-06-30 (Actual); Primary Completion 2015-12-13 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Chung, Principal Investigator — Eastern Cooperative Oncology Group
Locations (272):
- United States (272):
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Veteran's Administration Medical Center, Little Rock, Arkansas
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Saint Joseph Regional Medical Center, Lewiston, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer, Sandpoint, Idaho
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Saint Joseph Hospital, Chicago, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium Community Clinical Oncology Program, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Community Hospital, Niles, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro-Minnesota CCOP, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Phelps County Regional Medical Center, Rolla, Missouri
  - Saint John's Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Ozark Health Ventures LLC-Cancer Research for The Ozarks Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Billings Clinic, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Oncology Hematology West, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Oncology Hematology West PC, Omaha, Nebraska
  - Urology Cancer Center PC, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - New York Oncology Hematology PC - Albany, Albany, New York
  - New York Oncology Hematology PC -Albany Medical Center, Albany, New York
  - New York Oncology Hematology PC-Hudson, Hudson, New York
  - New York Oncology Hematology PC - Latham, Latham, New York
  - Orange Regional Medical Center, Middletown, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Oncology Hematology PC - Troy, Troy, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Southeastern Medical Oncology Center-Wilson, Wilson, North Carolina
  - Akron General Medical Center, Akron, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - University Pointe, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Western Oncology Research Consortium, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology at Evangelical Community Hospital, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Pottstown Memorial Medical Center, Pottstown, Pennsylvania
  - Geisinger Medical Oncology-Pottsville, Pottsville, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Wellmont Bristol Regional Medical Center, Bristol, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Johnson City, Johnson City, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Kingsport, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - University Medical Center Brackenridge, Austin, Texas
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Auburn Regional Medical Center, Auburn, Washington
  - Overlake Hospital Medical Center, Bellevue, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Saint John Medical Center, Longview, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - Capital Medical Center, Olympia, Washington
  - Good Samaritan Community Hospital, Puyallup, Washington
  - Allenmore Hospital, Tacoma, Washington
  - Northwest CCOP, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Multicare Health System, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - West Virginia University Charleston, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Riverview Hospital, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A (Afatinib) | Arm B (Placebo)
Started | 2 | 1
Completed | 0 | 0
Not Completed | 2 | 1
Not completed — Lack of Efficacy | 1 | 1
Not completed — Off-treatment reason not submitted | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Afatinib) | Arm B (Placebo) | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival (DFS)
Description: DFS is defined as the time from randomization to the earlier of disease recurrence, second primary cancer, or death without recurrence.
Time Frame: Assessed every 3 months for patients < 2 years from registration and every 6 months if patient is 2-3 years from registration and every 12 months if patient is 4-5 years from registration
Population: All randomized patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Afatinib) | Arm B (Placebo)
Number analyzed (Participants) | 2 | 1
months | NA [5.2 to NA] — The estimated median DFS was not available by definition in the survival setting. The upper limit of the 95% CI was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | NA [NA to NA] — Individual data could not be reported for patient privacy reasons as only 1 patient was enrolled in this arm.

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment.
Arm/Group | Arm A (Afatinib) | Arm B (Placebo)
Serious Adverse Events (participants affected / at risk) | 2/2 | 1/1
Other Adverse Events (participants affected / at risk) | 2/2 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Afatinib) (N=2) | Arm B (Placebo) (N=1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Confusion (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Afatinib) (N=2) | Arm B (Placebo) (N=1)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0
Mucositis oral (Gastrointestinal disorders) | 2 | 0
Lymphocyte count decreased (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 0
Spasticity (Musculoskeletal and connective tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Due to the small sample size, estimates on median DFS and 95% confidence intervals could be unreliable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less